CLINICAL TRIAL: NCT03797807
Title: Clinical and Radiographic Changes in Intrabony Defects Following Non-surgical vs. Surgical Minimally-invasive Periodontal Therapy. A Parallel Group, Single Centre, Examiner-blind, Non-inferiority Randomised Controlled Trial
Brief Title: Minimally-invasive Non-surgical and Surgical Periodontitis Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/LO/1956
Record Dates: First submitted 2018-12-19; First posted 2019-01-09 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MINST (Experimental): Minimally invasive non surgical treatment
  Interventions: Procedure: MINST
- MIST (Active Comparator): Minimally invasive surgical treatment
  Interventions: Procedure: MIST
- GTI + MINST (Active Comparator): Minimally invasive non surgical treatment + Geometric/Thermal Imaging (GTI subgroup)
  Interventions: Procedure: MINST; Diagnostic Test: GTI subgroup (Geometrical/Thermal Imaging)
- GTI + MIST (Active Comparator): Minimally invasive surgical treatment + Geometric/Thermal Imaging (GTI subgroup)
  Interventions: Procedure: MIST; Diagnostic Test: GTI subgroup (Geometrical/Thermal Imaging)

INTERVENTIONS:
Procedure: MINST — A non-surgical minimally invasive treatment protocol, named MINST, has been proposed for the treatment of periodontal intrabony defects, in order to minimize patient discomfort and maximize the healing potential
  Arms: GTI + MINST; MINST
Procedure: MIST — A minimally invasive surgical treatment protocol, named MIST, has been proposed for the treatment of periodontal intrabony defects, in order to minimize patient discomfort and maximize the healing potential
  Arms: GTI + MIST; MIST
Diagnostic Test: GTI subgroup (Geometrical/Thermal Imaging) — Geometrical/Thermal Imaging
  Arms: GTI + MINST; GTI + MIST

SUMMARY:
To compare the efficacy of a modified minimally-invasive non-surgical periodontal therapy (MINST) approach with a surgical approach (M-MIST) in determining bone and clinical attachment changes in intrabony defects

DETAILED DESCRIPTION:
Periodontal diseases are inflammatory conditions that affect the supporting apparatus of the teeth, including gingiva and alveolar bone. The bone loss resulting from periodontitis often is irregular and localised, giving onset to 'intrabony' or 'vertical defects' affecting one side of the tooth more than the other and more than on the neighbouring teeth. Periodontal intrabony defects have been associated with a higher risk of further progression and eventually tooth loss.

The treatment of periodontitis involves a non-specific reduction of the bacterial load below the gingival margin. This is achieved by oral hygiene instructions (OHI) and non-surgical periodontal therapy (NSPT), aimed at removing calculus and disrupting the plaque biofilm from the affected root surfaces. Intrabony defects are considered sites requiring therapy, often beyond NSPT. Decades ago, intrabony defects were treated with surgical elimination of the defect achieved by sacrificing the adjacent healthy supportive or non-supportive bone. More recently periodontal regenerative procedures have been advocated for deep intrabony defects, which are considered amenable for guided tissue regeneration. This technique results in regeneration of periodontal attachment measurable histologically and radiographically and measurable clinically. However, this is associated with potential morbidity and high costs due to the use of bone graft and barrier materials and is not always predictable. The more recent introduction of minimally-invasive surgical therapy (MIST), modified-MIST (M-MIST) and single-flap approach suggested that the use of biomaterials may not be so crucial for obtaining periodontal regeneration.

Retrospective studies from the investigator's group have shown that minimally invasive non-surgical periodontal treatment of intrabony defects results in clinical improvements (measured as PPD reductions and clinical attachment level-CAL- gain) but also in bone fill of the bony defects, measurable radiographically. The extent of the radiographic resolution of the defect was positively associated with initial defect depth and use of adjunctive antibiotics, while smoking seemed to negatively influence this outcome. A non-surgical minimally-invasive treatment protocol, named MINST, has been proposed along these principles. A more recent retrospective analysis has revealed a reduction in bony defect of nearly 3 mm for cases treated with minimally-invasive non-surgical therapy. The effect of MINST may be mediated by improved blood flow and stable blood clot in the intrabony defect. However, very few studies have been published on MINST and no data are available on the comparison between MINST and MIST.

This is a parallel group, single centre, examiner-blind, non-inferiority randomized controlled trial to compare the effect of a modified minimally-invasive non-surgical therapy (MINST) approach to minimally invasive surgical treatment (MIST) in the healing of periodontal intrabony defects in 66 patients with periodontitis .

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-70
2. Diagnosis of 'Periodontitis' stage III or IV (grades A to C)
3. Presence of ≥1 'intrabony defect' (PPD, >5 mm with intrabony defect depth ≥3mm at screening radiograph),
4. Signed informed consent. -

Exclusion Criteria:

1. Smoking (current or in past 5 years) including e-cigarettes/vaping 2. Medical history including diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases 3. History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures 4. Antiinflammatory or anticoagulant therapy during the month preceding the baseline exam 5. Systemic antibiotic therapy during the 3 months preceding the baseline exam 6. History of alcohol or drug abuse, 7. Self-reported pregnancy or lactation 8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that according to the investigator may increase the risk associated with trial participation, 9. Periodontal treatment to the study site within the last 12 months (excluding not-extensive subgingival debridement as judged by the examining clinician).

-

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic whole defect depth change | 9 months
  Radiographic whole defect depth change in millimeters at 9 months [considered a surrogate measure evaluating the entire regenerative process including bone, cementum and periodontal ligament

OTHER OUTCOMES:
Probing Pocket Depth (PPD) change | Up to 15 months
  Probing Pocket Depth (PPD) change (in mm)
Clinical Attachment Level (CAL) gain change | Up to 15 months
  Clinical Attachment Level (CAL) gain change (in mm)
Markers and growth factors in gingival crevicular fluid (GCF) | Up to 15 months
  Levels of inflammatory markers and growth factors in gingival crevicular fluid (GCF). Specifically, markers related with the healing of epithelium, connective tissue, bone and related to inflammatory/host responses will be examined.
Bacterial detection | Up to 15 months
  Bacterial detection associated with presence of intrabony defects
Gingival inflammation and healing | Up to 15 months
  Gingival inflammation and healing (as measured by geometric/thermal stereophotogrammetry imaging in the 'GTI sub-study')
Self administered OIDP (oral impact on daily performances index) | Up to 9 months
  We will utilize the oral impact on daily performances index (OIDP) to evaluate health and treatment outcomes. The OIDP focuses on the impact that the conditions of the teeth and mouth have on the physical/functional, psychological and social well-being of the person. Particularly, it assesses the impact of oral conditions on basic daily life activities and behaviours (eating, speaking, cleaning teeth, and going out, relaxing, smiling, major work or role, emotional stability, social contact). For each performance, both the frequency and severity of oral impacts are assessed. The overall OIDP score ranges from 0 to 100, with higher scores indicating worse quality of life.
Global ratings on health and quality of life with Visual Analogue Scale (VAS) | Up to 9 months
  The VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Global ratings on health and quality of life with a question "How would you rate the quality of your life" | Up to 9 months
  The responses will be scored on a six-point scale as:
  1. Excellent
  2. Very good
  3. Good
  4. Fair
  5. Poor
  6. Very poor

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, PhD, Principal Investigator — Barts & The London School of Medicine & Dentistry, QMUL
Locations (1):
- Barts and The London Dental Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papapanou PN, Tonetti MS. Diagnosis and epidemiology of periodontal osseous lesions. Periodontol 2000. 2000 Feb;22:8-21. doi: 10.1034/j.1600-0757.2000.2220102.x. No abstract available. PMID 11276518
- [Background] Papapanou PN, Wennstrom JL. The angular bony defect as indicator of further alveolar bone loss. J Clin Periodontol. 1991 May;18(5):317-22. doi: 10.1111/j.1600-051x.1991.tb00435.x. PMID 2066446
- [Background] Heitz-Mayfield LJ, Trombelli L, Heitz F, Needleman I, Moles D. A systematic review of the effect of surgical debridement vs non-surgical debridement for the treatment of chronic periodontitis. J Clin Periodontol. 2002;29 Suppl 3:92-102; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.5.x. PMID 12787211
- [Background] Nyman S, Lindhe J, Karring T, Rylander H. New attachment following surgical treatment of human periodontal disease. J Clin Periodontol. 1982 Jul;9(4):290-6. doi: 10.1111/j.1600-051x.1982.tb02095.x. PMID 6964676
- [Background] Cortellini P, Tonetti MS. Focus on intrabony defects: guided tissue regeneration. Periodontol 2000. 2000 Feb;22:104-32. doi: 10.1034/j.1600-0757.2000.2220108.x. No abstract available. PMID 11276509
- [Background] Needleman IG, Worthington HV, Giedrys-Leeper E, Tucker RJ. Guided tissue regeneration for periodontal infra-bony defects. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD001724. doi: 10.1002/14651858.CD001724.pub2. PMID 16625546
- [Background] Trombelli L, Farina R, Franceschetti G, Calura G. Single-flap approach with buccal access in periodontal reconstructive procedures. J Periodontol. 2009 Feb;80(2):353-60. doi: 10.1902/jop.2009.080420. PMID 19186978
- [Background] Cortellini P, Tonetti MS. Clinical and radiographic outcomes of the modified minimally invasive surgical technique with and without regenerative materials: a randomized-controlled trial in intra-bony defects. J Clin Periodontol. 2011 Apr;38(4):365-73. doi: 10.1111/j.1600-051X.2011.01705.x. Epub 2011 Feb 8. PMID 21303402
- [Background] Nibali L, Pometti D, Tu YK, Donos N. Clinical and radiographic outcomes following non-surgical therapy of periodontal infrabony defects: a retrospective study. J Clin Periodontol. 2011 Jan;38(1):50-7. doi: 10.1111/j.1600-051X.2010.01648.x. Epub 2010 Nov 22. PMID 21091528
- [Background] Ribeiro FV, Casarin RC, Palma MA, Junior FH, Sallum EA, Casati MZ. Clinical and patient-centered outcomes after minimally invasive non-surgical or surgical approaches for the treatment of intrabony defects: a randomized clinical trial. J Periodontol. 2011 Sep;82(9):1256-66. doi: 10.1902/jop.2011.100680. Epub 2011 Feb 2. PMID 21284549
- [Background] Nibali L, Pometti D, Chen TT, Tu YK. Minimally invasive non-surgical approach for the treatment of periodontal intrabony defects: a retrospective analysis. J Clin Periodontol. 2015 Sep;42(9):853-859. doi: 10.1111/jcpe.12443. Epub 2015 Sep 29. PMID 26257238
- [Derived] Nibali L, Koidou V, Salomone S, Hamborg T, Allaker R, Ezra R, Zou L, Tsakos G, Gkranias N, Donos N. Minimally invasive non-surgical vs. surgical approach for periodontal intrabony defects: a randomised controlled trial. Trials. 2019 Jul 27;20(1):461. doi: 10.1186/s13063-019-3544-8. PMID 31351492